CLINICAL TRIAL: NCT00345332
Title: A Multi-Center, Double-Blind, Randomized, Placebo-Controlled Trial of Botox for Severe Refractory Urge Urinary Incontinence
Brief Title: A Multi-Center Trial of Botox for Severe Urge Urinary Incontinence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 12299
Record Dates: First submitted 2006-06-27; First posted 2006-06-28 (Estimated); Results first posted 2017-07-11 (Actual); Last update posted 2017-07-11 (Actual); Status verified 2017-06

CONDITIONS: Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- 2 (Experimental): Botox
  Interventions: Drug: Botox

INTERVENTIONS:
Drug: Botox — Injected
  Arms: 2
Drug: Placebo — Injected
  Arms: 1

SUMMARY:
The purpose of the study is to determine how effective Botox is in reducing the amount of urine leaked and which dose of Botox is more effective and safe in those who have urinary urge incontinence.

DETAILED DESCRIPTION:
A multi-center clinical trial of Botulinum-A Toxin (Botox) for refractory urge incontinence.

ELIGIBILITY:
Inclusion Criteria:

* Female subjects 21-90 years of age
* subjects has urinary incontinence on 3 day bladder diary
* subject has severe incontinence
* urine dipstick or urine culture negative for urinary tract infection
* cystometrogram without stress urinary leakage
* must have failed at least one anti-cholinergic medication
* negative urine pregnancy test on day of administration of study medication

Exclusion Criteria:

* history of carcinoma of the bladder
* presence of foreign body in the bladder, cystitis or other correctable etiology for Urge Urinary Incontinance
* gross fecal incontinence
* known allergy to sulfa or ciprofloxacin or to lidocaine
* any medical condition that may put the subject at increased risk with exposure to Botox
* females who are pregnant, breast-feeding, or planning a pregnancy during the study or who are of child-bearing potential
* known allergy to any of the components in the study medication
* prior documented resistance to Botox
* evidence of recent alcohol or drug abuse
* concurrent participation in another investigational drug or device study within 30 days

Ages: 21 Years to 90 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2005-10; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael K Flynn, MD, Principal Investigator — University of Rochester
Locations (3):
- United States (3):
  - University of California at Davis, Sacramento, California
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Duke University Medical Center, Durham, North Carolina

REFERENCES:
- [Result] Flynn MK, Webster GD, Amundsen CL. The effect of botulinum-A toxin on patients with severe urge urinary incontinence. J Urol. 2004 Dec;172(6 Pt 1):2316-20. doi: 10.1097/01.ju.0000143889.00681.3f. PMID 15538257

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo Group: 6 cc of saline was administered into the detrusor along the bladder base. We injected 0.5 ccs at each injection site.
- Botox Group: Botox (BTX) was administered into the detrusor along the bladder base. BTX was reconstituted in 6 ccs of preservative free saline according to manufacturers instructions. We injected 0.5 ccs at each injection site.
Period: Overall Study
Arm/Group | Placebo Group | Botox Group
Started | 11 | 20
Completed | 11 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Botox Group: BTX was administered into the detrusor along the bladder base. BTX was reconstituted in 6 ccs of preservative free saline according to manufacturers instructions. We injected 0.5 ccs at each injection site.
- Total: Total of all reporting groups
Arm/Group | Placebo Group | Botox Group | Total
Number analyzed (Participants) | 11 | 20 | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.45 (12.85) | 65.15 (10.83) | 65.97 (11.55)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 20 | 31
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 11 | 20 | 31

OUTCOME MEASURES:

1. Primary Outcome: Incontinent Episodes Per Day
Description: The number of incontinence episodes per day was recorded by each participant in a diary. All incontinence episodes were counted when calculating episodes per day at each time point.
Time Frame: week 13
Measure: Geometric Least Squares Mean (Standard Error); unit: incontinence episodes per day
Arm/Group | Placebo Group | Botox Group
Number analyzed (Participants) | 11 | 20
incontinence episodes per day | 7.34 (1.07) | 3.90 (0.75)
Statistical Analysis 1: Comparison: Botox Group; Test type: Superiority or Other; p < 0.01, ANOVA

2. Secondary Outcome: Number of Incontinence Pads Used Per Day
Description: The number of incontinence pads used per day per day was recorded by each participant in a diary.
Time Frame: week 13
Measure: Geometric Least Squares Mean (Standard Error); unit: pads per day
Arm/Group | Placebo Group | Botox Group
Number analyzed (Participants) | 11 | 20
pads per day | 5.18 (0.92) | 3.13 (0.66)
Statistical Analysis 1: Comparison: Botox Group; Test type: Superiority or Other; p < 0.01, ANOVA

ADVERSE EVENTS:
Arm/Group | Placebo Group | Botox Group
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/20
Other Adverse Events (participants affected / at risk) | 3/11 | 11/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Group (N=11) | Botox Group (N=20)
urinary tract infection (Infections and infestations) | 3 | 11
post void retention volumes > 200cc (Renal and urinary disorders) | 0 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No